CLINICAL TRIAL: NCT01869478
Title: Endovascular Arterial Reperfusion vs. Intravenous ThromboLYsis for Acute Ischemic Stroke (EARLY): A Randomized Pilot Study of Ultra-early (<2 Hours) and Early (2-4.5 Hours) Reperfusion Therapy
Brief Title: Feasibility Study of IV Recombinant Tissue Plasminogen Activator (rtPA) vs. Primary Endovascular Therapy for Acute Ischemic Stroke
Acronym: EARLY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin M. Barrett, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-002496
Record Dates: First submitted 2013-06-01; First posted 2013-06-05 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Thrombolysis (Active Comparator): 0.9mg/kg intravenous rt-PA (max dose 90mg) - 10% administered as a bolus over 1 minute and the remainder infused over 60 minutes.
  Interventions: Drug: Intravenous Thrombolysis
- Endovascular Arterial Reperfusion (Active Comparator): Therapeutic options will include mechanical thrombectomy/clot disruption (Penumbra aspiration system, Solitaire device, and/or Reflex catheter) and/or intracranial stent deployment.
  Interventions: Device: Endovascular Arterial Reperfusion

INTERVENTIONS:
Drug: Intravenous Thrombolysis
  Other Names: Altelplase, rtPA
  Arms: Intravenous Thrombolysis
Device: Endovascular Arterial Reperfusion
  Other Names: Penumbra, Solitaire
  Arms: Endovascular Arterial Reperfusion

SUMMARY:
This pilot trial will be the first step toward direct comparison of delivery of endovascular reperfusion therapy to intravenous recombinant tissue plasminogen activator (rt-PA) in a time-to-treatment framework shown as most effective by the NINDS rt-PA Stroke Trial. A randomized trial is justified for the following reasons: 1) The high rate of death and disability associated with ischemic stroke despite treatment with intravenous rt-PA mandates critical analysis of alternate therapies with therapeutic potential, 2) endovascular treatment for acute ischemic stroke is expanding in North America without compelling evidence of safety and efficacy from well-designed clinical trials, 3) critical cost-effectiveness analysis cannot be done without acquiring pertinent outcomes data from controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Definite or probable ischemic stroke
* CT angiographic (CTA) evidence of intracranial vascular occlusion (internal carotid, middle cerebral - M1 or M2 divisions, anterior cerebral, posterior cerebral, or basilar artery) within 3.5 hours of symptom onset
* Able to receive assigned treatment within 4.5 hours of symptom onset
* Written informed consent from patient or surrogate, if unable to provide consent

Exclusion Criteria:

* CT evidence of early infarction in >1/3 of middle cerebral artery distribution
* Blood pressure > 185/110 mmHg refractory to anti-hypertensive therapy
* History of intracranial hemorrhage
* History of ischemic stroke within past 3 months
* History of major surgical procedure within past 14 days
* Gastrointestinal or genitourinary bleeding within past 14 days
* Glucose <50 or >400mg/dL
* Platelet count <100,000
* International normalized ratio (INR) ≥ 1.7
* Known history of bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Barrett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Thrombolysis | Endovascular Arterial Reperfusion
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Thrombolysis | Endovascular Arterial Reperfusion | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recanalization Rate of Primary Intracranial Occlusion
Description: The degree of recanalization (none, partial, complete) will be assessed in a blinded fashion on the 24-hour computed tomographic angiogram (CTA).
Time Frame: 24 hours
Population: Only one participant was enrolled, so data analysis was not possible.
Arm/Group | Intravenous Thrombolysis | Endovascular Arterial Reperfusion
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Score on Modified Rankin Scale at 90 Days
Description: Functional outcome at 90-days will be assessed with the modified Rankin Scale (mRS). The Modified Rankin Scale was completed by the physician; it is a 7 point scale rating any limitations in the study subject's social role. The scale ranges from 0 (no symptoms/disability) to 6 (death).
Time Frame: 90 days
Population: Only one participant was enrolled, so data analysis was not possible.
Arm/Group | Intravenous Thrombolysis | Endovascular Arterial Reperfusion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Thrombolysis | Endovascular Arterial Reperfusion
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
This study was terminated due to difficulty in recruiting subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes